CLINICAL TRIAL: NCT06820203
Title: Comparison Between Premixed, Sequential and Manually Mixed Administration of Intrathecal Fentanyl and Bupivacaine in Cesarean Section: A Randomized Controlled Study
Brief Title: Premixed, Sequential and Manually Mixed Administration of Intrathecal Fentanyl and Bupivacaine in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1048/1/25
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Premixed; Sequential; Manually Mixed; Intrathecal; Fentanyl; Bupivacaine; Cesarean Section
MeSH Terms: interventions — Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Premixed group (Experimental): Patients will receive premixed intrathecal fentanyl and bupivacaine in the same syringe.
  Interventions: Drug: Fentanyl and Bupivacaine
- Sequential group (Experimental): Patients will receive intrathecal fentanyl and bupivacaine in separate syringes.
  Interventions: Drug: Fentanyl and Bupivacaine
- Manual mixed group (Active Comparator): Patients will receive manually mixed intrathecal fentanyl and bupivacaine in the same syringe.
  Interventions: Drug: Fentanyl and Bupivacaine

INTERVENTIONS:
Drug: Fentanyl and Bupivacaine — Patients will receive premixed intrathecal fentanyl and bupivacaine in the same syringe.
  Arms: Premixed group
Drug: Fentanyl and Bupivacaine — Patients will receive intrathecal fentanyl and bupivacaine in separate syringes.
  Arms: Sequential group
Drug: Fentanyl and Bupivacaine — Patients will receive manually mixed intrathecal fentanyl and bupivacaine in the same syringe.
  Arms: Manual mixed group

SUMMARY:
This study aims to distinguish between premixed, sequential, and manually mixed administration of intrathecal fentanyl and bupivacaine in cesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is a lifesaving procedure when there is both maternal and fetal problems. The rate of CS increases dramatically from time to time. Regional anesthesia techniques are highly preferred for CS compared to general anesthesia.

Coadministration of intrathecal opioids and local anesthetics (LAs) have been found to produce a potent intra and postoperative analgesic synergism without further depression of efferent sympathetic activity, hence results in less adverse hemodynamic effects, even with sub-therapeutic doses of LAs.

Fentanyl has been considered the intrathecal LAs adjuvant of choice owing to its potency, fast onset and short duration of action, and lower incidence of respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* Height between 150 to175 cm.
* Body mass index (BMI) between 18.5 and 30 kg/m2.
* American Society of Anesthesiology (ASA) physical status II.
* Scheduled for cesarean section under spinal anesthesia.

Exclusion Criteria:

* Pre-operation hypotension and bradycardia.
* Preeclampsia.
* Multiple pregnancy and macrosomia.
* Complete or partial failed spinal.
* Patients with skin infections at the site of injection.
* Patients with coagulation disorders.
* Patients with spinal deformities.
* Patients having regional nerve block other than spinal anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing cesarean section
Enrollment: 90 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of pethidine administrated).

SECONDARY OUTCOMES:
Total analgesic consumption | 24 hours postoperatively
  The total amount of analgesic the patient will be given within 24 h after spinal anesthesia
Degree of pain | 24 hours postoperatively
  The degree of pain will be assessed using the numerical rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at 0, 2, 4, 6, 8, 12, 18, and 24h postoperatively.
Onset of motor block | Intraoperatively
  onset of motor block (defined as the time from giving spinal anesthesia until a modified Bromage score of 3 was reached). The modified Bromage scale [0: No motor block, 1: Unable to raise an extended leg (able to flex the knee), 2: Unable to flex the knee (able to move the foot only), 3: Unable to flex the ankle (unable to move the foot or knee)]
Duration of motor block | Intraoperatively
  Duration of motor block (defined as the time from the onset of motor blockade until complete recovery, indicated by a Bromage score of 0) will be recorded
Onset of sensory block | Intraoperatively
  Onset of sensory block (time elapsed from the end of spinal injection to absence of pinprick sensation at T10 dermatome).
Duration of sensory block | Intraoperatively
  Duration of sensory block (The time till achieving T10 sensory level in addition to the maximum block height) will be noted and recorded.
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as bradycardia, hypotension, nausea, Pruritus, shivering, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.